CLINICAL TRIAL: NCT00805194
Title: Multicentre, Randomised, Double-blind, Phase III Trial to Investigate the Efficacy and Safety of Oral BIBF 1120 Plus Standard Docetaxel Therapy Compared to Placebo Plus Standard Docetaxel Therapy in Patients With Stage IIIB/IV or Recurrent Non Small Cell Lung Cancer After Failure of First Line Chemotherapy
Brief Title: LUME-Lung 1: BIBF 1120 Plus Docetaxel as Compared to Placebo Plus Docetaxel in 2nd Line Non Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1199.13; 2007-004803-36 (EudraCT Number)
Record Dates: First submitted 2008-12-08; First posted 2008-12-09 (Estimated); Results first posted 2014-12-01 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel; nintedanib

ARMS (2):
- BIBF 1120 plus docetaxel (Experimental): BIBF 1120 2 times daily along with standard therapy of docetaxel
  Interventions: Drug: BIBF 1120 plus docetaxel
- Placebo plus docetaxel (Placebo Comparator): Placebo matching BIBF 1120 2 times daily along with standard therapy of docetaxel
  Interventions: Drug: placebo plus docetaxel

INTERVENTIONS:
Drug: placebo plus docetaxel — placebo matching BIBF 1120 2 times daily along with standard therapy of docetaxel
  Arms: Placebo plus docetaxel
Drug: BIBF 1120 plus docetaxel — BIBF 1120 2 times daily along with standard therapy of docetaxel
  Arms: BIBF 1120 plus docetaxel

SUMMARY:
The present trial will be performed to evaluate whether BIBF 1120 in combination with standard therapy of docetaxel in patients with stage IIIB/IV or recurrent NSCLC is more effective as compared to placebo in combination with standard therapy of docetaxel. A secondary aim is to obtain safety information as well as information on quality of life of patients treated with BIBF 1120 in combination to standard therapy with docetaxel. In addition, blood will be collected for pharmacokinetic analysis.

ELIGIBILITY:
Inclusion criteria:

* male or female patient aged 18 years or older;
* histologically or cytologically confirmed, locally advanced and/or metastatic NSCLC of stage IIIB or IV or recurrent NSCLC;
* relapse or failure of one first line prior chemotherapy;
* at least one target tumour lesion that has not been irradiated within the past three months and that can accurately be measured ;
* life expectancy of at least three months;
* Eastern Cooperative Oncology group (ECOG) score of 0 or 1;
* patient has given written informed consent

Exclusion criteria:

* more than one prior chemotherapy regimen for advanced and/or metastatic or recurrent NSCLC;
* more than one chemotherapy treatment regimen (either neoadjuvant or adjuvant or neoadjuvant plus adjuvant) prior to first line chemotherapy;
* previous therapy with other VEGFR inhibitors (other than bevacizumab) or docetaxel for treatment of NSCLC;
* persistence of clinically relevant therapy related toxicities from previous chemotherapy and/or radiotherapy;
* treatment with other investigational drugs or other anti-cancer therapy or treatment in another clinical trial within the past four weeks before start of - therapy or concomitantly with this trial ;
* radiotherapy (except extremities and brain) within the past three months prior to baseline imaging;
* active brain metastases or leptomeningeal disease;
* radiographic evidence of cavitary or necrotic tumours;
* centrally located tumours with radiographic evidence (CT or MRI) of local invasion of major blood vessels;
* history of clinically significant haemoptysis within the past 3 months;
* therapeutic anticoagulation (except low dose heparin) or antiplatelet therapy;
* history of major thrombotic or clinically relevant major bleeding event in the past 6 months;
* known inherited predisposition to bleeding or thrombosis;
* significant cardiovascular diseases ;
* inadequate safety laboratory parameters;
* significant weight loss (> 10 %) within the past 6 weeks;
* current peripheral neuropathy greater than CTCAE grade 2 except due to trauma;
* preexisting ascites and/or clinically significant pleural effusion;
* major injuries and/or surgery within the past ten days prior to randomisation with incomplete wound healing;
* serious infections requiring systemic antibiotic therapy;
* decompensated diabetes mellitus or other contraindication to high dose corticosteroid therapy;
* gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug;
* active or chronic hepatitis C and/or B infection;
* serious illness or concomitant non-oncological disease or laboratory abnormality that may increase the risk associated with study participation or study drug administration;
* patients who are sexually active and unwilling to use a medically acceptable method of contraception during the trial and for at least twelve months after end of active therapy;
* pregnancy or breast feeding;
* psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule;
* patients unable to comply with the protocol;
* active alcohol or drug abuse;
* other malignancy within the past three years other than basal cell skin cancer, or carcinoma in situ of the cervix;
* any contraindications for therapy with docetaxel;
* history of severe hypersensitivity reactions to docetaxel or other drugs formulated with polysorbate 80 (Tween 80);
* hypersensitivity to BIBF 1120 and/or the excipients of the trial drugs;
* hypersensitivity to contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1314 (Actual)
Dates: Start 2008-12-03 (Actual); Primary Completion 2010-11-02 (Actual); Study Completion 2017-11-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (210):
- Austria (3):
  - LKH-Univ. Hospital Graz, Graz
  - KH St. Vinzenz, Zams, Int. Abtlg., Kufstein
  - AKH d. Stadt Linz, Pulmologie, Linz
- Belarus (7):
  - Bobruisk Inter-distict, Babruysk
  - Brest Regional Clinical, Brest Region
  - Gomel Regional Clinical, Homyel
  - Public Health Inst. Minsk City Clinical Oncology Dispensary, Minsk
  - Scientific Research Minsk, Minsk Region
  - Mogilov Regional Oncological Dispensary, Mogilev
  - Vitebsk Regional Clinical Oncology Dispensary, Vitebsk
- Belgium (2):
  - Centre Hospitalier Universitaire de Liège, Liège
  - Liège - HOSP CHR de la Citadelle, Liège
- Bulgaria (6):
  - Multiprofile Hospital for Active Treatment, Gabrovo
  - Univ.Multiprofile Hospital "Dr. Georgy Stranski" EAD, Pleven, Pleven
  - District Oncology Dispensary Plovdiv, Plovdiv
  - Interdistrict Oncology Dispensary, Ruse, Rousse
  - District Oncology Dispensary Shumen, Shumen
  - Specialized Hospital for Active Treatment in Oncolcogy, Sofia
- China (20):
  - 307 Hospital of PLA, Beijing
  - Jilin Province Cancer Hospital, Changchun
  - First Hospital of Jilin University, Changchun
  - West China Hospital, Chengdu
  - Southwest Hospital, Chongqing
  - First Affiliated Hospital of Dalian Medical University, Dalian
  - The Second Affiliated Hospital of Dalian Medical University, Dalian
  - Fujian Provincial Tumor Hospital, Fujian
  - Sun Yat-Sen University Cancer Center, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - Sir Run Run Shaw Hospital, Hangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - The Third Affiliated Hospital of Harbin Medical University, Harbin
  - the 81th Hospital of PLA, Nanjing
  - Jiangsu Cancer Hospital, Nanjing
  - Shanghai Chest Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
  - Shanghai Pulmonary Hospital, Shanghai
  - Tongji Hospital, Tongji University, Wuhan
  - Zhongshan Hospital Fudan University, Xuhui Area, Shanghai
- Croatia (2):
  - Clinical Hospital Centar Sestre Milosrdnice, Zagreb
  - UHC Zagreb, Zagreb
- Czechia (5):
  - University Hospital Brno, Brno
  - St. Anna Hospital, 2nd Internal Department, Brno
  - District Hospital Liberec, Liberec
  - Institut onkologie a rehabilitace Na Plesi s.r.o., Nová Ves pod Pleší
  - District Hospital Pribram, Oncology Centrum, Příbram
- Denmark (2):
  - Herlev Hospital, Herlev
  - Odense Universitetshospital, Odense C
- France (8):
  - HOP Croix Rousse, Pneumo, Lyon, Lyon
  - INS Paoli-Calmettes, Marseille
  - HOP Lyon Sud, Pierre-Bénite
  - CHU de Rouen - Hôpital de Bois Guillaume, Rouen
  - HOP Nord Laënnec, Saint-Herblain
  - Oncology Institute of the Loire, Saint-Priest-en-Jarez
  - HOP Civil, Strasbourg
  - Sainte Anne Training hospital for the armies, Toulon
- Georgia (3):
  - Amtel Hospital first Clinical LLC, Tbilisi
  - National Centre of Oncology, Tbilisi
  - Chemotherapy & Immunotherapy Clinic 'Medulla', Tbilisi, Tbilisi
- Germany (30):
  - Gemeinschaftspraxis Dr. Brudler / Dr. Heinrich, Augsburg, Augsburg
  - Zentralklinik Bad Berka GmbH, Bad Berka
  - Universitätsklinikum Benjamin Franklin, Berlin, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - Evangelische Lungenklinik Berlin, Buch
  - Gemeinschaftspraxis für Hämatologie und Onkologie, Köln, Cologne
  - Universitätsklinikum Frankfurt, Frankfurt
  - Krankenhaus Nordwest, Frankfurt, Frankfurt am Main
  - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Asklepios Fachkliniken München-Gauting, Gauting
  - Pneumologisches Forschungsinstitut an der LungenClinic Grosshansdorf GmbH, Großhansdorf
  - Krankenhaus Martha-Maria Halle-Dölau gGmbH, Halle
  - Allgemeines Krankenhaus Harburg, 21075 Hamburg, Hamburg
  - Universitätsklinikum Heidelberg, Heidelberg
  - Klinikum Kassel GmbH, Kassel
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - POIS Leipzig GbR, Leipzig
  - Klinik, Löwenstein, Löwenstein
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Lübeck
  - Katholisches Klinikum St. Hildegardiskrankenhaus, Mainz, Mainz
  - Universitätsmedizin der Johannes Gutenberg-Universität Mainz, Mainz
  - Universitätsklinik links der Isar, München, Ziemssenstr. 1, München
  - Klinikum rechts der Isar der Technischen Universität München, München
  - Städt. Krankenhaus, München-Bogenhausen, München
  - Pius-Hospital, Oldenburg, Oldenburg
  - Universitätsklinikum Tübingen, Tübingen
  - Helios Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
  - Evangelisches Krankenhaus, Witten, Witten
- Greece (5):
  - Athens Hospital of Chest Diseasea "SOTIRIA", Athens
  - University Hospital of Heraklion, University Pulmonology Cl, Heraklio
  - Iaso General Hospital, Holargos, Athens
  - Papageorgiou Hospital, 1st Cardiological Cl., Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki
- India (19):
  - Vedanta Institute of Medical Sciences, Ahmedabad
  - KIDWAI memoraial Institute of oncology, Bangalore
  - Rajalakshmi Multispeciality Hospital, Bangalore
  - Jawaharlal Nehru Cancer Hospital & Research Centre, Bhopal, M.P.
  - Apollo Hospital, Chennai
  - Birla Cancer Centre, Jaipur
  - Bhagwan Mahaveer Cancer Hospital & Research Center, Jawahar, Jaipur
  - SEAROC cancer center,S.K.soni Hospital, Jaipur, Rajasthan
  - B. P .Poddar Hospital & Medical Research Ltd., Kolkata, West Bengal
  - Kasturba Medical College and Hospital, Mangalore
  - Tata Memorial Centre, Mumbai
  - Shatabdi Superspeciality Hospital, Nashik
  - Sir Gangaram Hospital, New Delhi
  - Indraprastha Apollo Hospitals, New Delhi
  - Rajiv Gandhi Cancer Institute and Research Centre, New Delhi
  - Jehangir Hospital Oncology Department, Pune, Maharahtra
  - Regional Cancer Center, Trivandrum, Kerala
  - City Cancer Centre, Cancer Hospital & Research, Vijayawada
  - King George Hospital, Visakhapatnam
- Israel (6):
  - E. Wolfson Medical Center, Holon 58100, Holon
  - Hadassah Medical Center, Ein-Karem, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Sourasky Medical Center, Tel Aviv
  - The Chaim Sheba Medical Center Tel Hashomer, Tel Litwinsky
  - Assaf Harofe Medical Center, Ẕerifin
- Italy (11):
  - Az. Ospedaliere Umberto I di Ancona, Ancona
  - Centro di riferimento Oncologico, Aviano
  - Policlinico S. Orsola Malpighi, Bologna
  - Fond. Poliambulanza Istituto, Brescia
  - Azienda Ospedaliera Careggi, Florence
  - Ospedale Civile, Ivrea (TO)
  - Istituto Scientifico Romagnolo, Meldola
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Sanitaria Ospedale S. Luigi Gonzaga, Orbassano
  - Fondazione Salvatore Maugeri, Pavia
  - Ospedale S.Maria della Misericordia, AO di Perugia, Perugia
- Lithuania (3):
  - Hospital of Lithuanian Univ.of HealthSciences Kauno Klinikos, Kaunas
  - Siauliu ligonine, Siauliai, Šiauliai
  - Vilniaus Universiteto, Vilnius
- Poland (9):
  - Pulmonology Center in Bydgoszcz, Bydgoszcz
  - Regional Complex Hospital, Elblag
  - Institute of Tuberculosis & Pulmonology, III. Dept., Olsztyn, Olsztyn
  - Mazowieckiego Centrum, Otwock
  - Greater PL Cent.Pulmo.&Thor.Surg.Eugenia&Janusz Zeyland, Poznan
  - Independent Public Hospital in Suwalki, Suwałki
  - Specialist Hospital, Szczecin-Zdunowo, Szczecin
  - Regional Specialist Hospital, Słupsk
  - Onco.Cent. - Instit. of Maria Sklodowskiej-Curie, Warsaw
- Portugal (7):
  - IPO Porto Francisco Gentil, EPE, Coimbra
  - IPO Lisboa Francisco Gentil, EPE, Lisbon
  - CHLN, EPE - Hospital de Santa Maria, Lisbon
  - IPO Porto Francisco Gentil, EPE, Porto
  - Centro Hospitalar São João,EPE, Porto
  - CHS, EPE - Hospital de São Bernardo, Setúbal
  - Centro Hospitalar de Vila Nova de Gaia, Vila Nova de Gaia
- Romania (10):
  - Baia Mare Emergency County Hospital, Baia Mare
  - Spitalul Clinic Judetean de Urgenta Brasov, Brasov
  - Institute of Oncology 'Prof. Dr. Alexandru Trestioreanu', Bucharest
  - Institutul Oncologic "Prof. Dr. Ion Chiricuta", Cluj-Napoca
  - County Hospital "Dr. Alex Simionescu", Hunedoara
  - Centrul de Oncologie Medicala, Iași
  - Emergency Clinical County Hospital "Sf Spiridon", Iasi, Iași
  - Onesti County Hospital, Onești
  - Emergency County Hospital "Sf.loan cel Nou", Suceava
  - Oncomed SRL, Timișoara
- Russia (15):
  - SBIH of Arkhangelsk reg. "Arkhangelsk Clin. Onc. Dispensary", Arkhangelsk
  - GLPU Cheliabinsky, Chelyabinsk
  - GUZ Irkutsk Regional Oncology Dispensary, Irkutsk
  - St.Auton.Heal.Inst."Rep.Clin.Onc.Disp.of MoH of Rep. Tatarstan", Kazan'
  - RBIH "Kursk regional clinical oncology dispensary", Kursk
  - GUZ Regional Oncology Dispensary, Magnitogorsk, Magnitogorsk
  - FSBI "N.N Blokhin Med.Res.Cent.Onc."MoH of RF, Moscow
  - SBIH of Stavropol territory "Pyatigorsk Oncol. Dispensary", Pyatigorsk
  - GUZ "Regional Clinical Oncology Dispensary", Ryazan
  - GUZ Leningradskaya Regional Clin. Hospital, St. Petersburg, Saint Petersburg
  - 1stPavlov St.Med.Univ.St.-Petersburg Res.Inst., Saint Petersburg
  - SPb SBIH "City Clinical Oncological Dispensary", Saint Petersburg
  - FSBI "N.N. Petrov National Medical Research Center of Oncology" of MoH of RF, Saint Petersburg
  - GUZ "Oncological Dispesary #2", Sochi
  - GUZ Sverdlovsky Regional Oncology Dispensary, Yekaterinburg
- Faculty Hospital Trnava, Trnava, Slovakia
- South Africa (7):
  - GVI oncology Medi Clinic, Cape Town
  - Parklands Hospital, Durban
  - WCR CMJAH Clinical Trial Site, Johannesburg
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Langenhoven Drive Oncology Centre, Port Elizabeth
  - Pretoria Academic Hospital, Pretoria
  - Wilgers oncology, Pretoria
- South Korea (3):
  - Gachon University Gil Medical Center, Incheon
  - VHS Medical Center, Seoul
  - The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul
- Spain (8):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitario de Elche, Elche
  - Hospital Jerez de la Frontera, Jerez de La Frontera-Cádiz
  - Hospital La Princesa, Madrid
  - Hospital Quirónsalud Madrid, Pozuelo de Alarcón
  - Fundación Instituto Valenciano de Oncologia, Valencia
  - Servicio de Oncologia Radiotherapica, Valencia
  - Hospital Arnau de Vilanova, Valencia
- Switzerland (2):
  - Kantonsspital Aarau, Aarau
  - Kantonsspital Baden AG, Baden
- Ukraine (11):
  - Chernigiv Regional Oncology Centre, Chernihiv
  - Bukovynsk State Medical University, Chernivtsi
  - Chmelnytskyi Oblasnnyi Oncologichnyi Tsentr, Chmelnytskyi
  - City Clinical Hospital #4, Dnipropetrovsk State Medical Academy, Dnipropetrovsk
  - Donetsk Regional Antitumor Centre, Donetsk
  - Kharkiv Medical Acadamy of Postgraduate education, Kharkiv
  - Kryvorizskyi regional communal clinical oncology centre, Kryvyi Rig
  - Odesa Regional Oncological Centre, Odesa
  - Ternopil regional communal clinical oncology centre, Ternopil
  - Uzhgorod National University, Oncology Centre, Uzhhorod
  - Vinnytsia Regional Clinical Oncological Dispensary, Vinnytsia
- United Kingdom (5):
  - Royal Bournemouth and Christchurch Hospital, Bournemouth
  - Bristol Haematology & Onc. Ctr, Bristol
  - Broomfield Hospital, Chelmsford
  - Wythenshawe Hospital, Manchester
  - Poole Hospital, Poole

REFERENCES:
- [Derived] Gottfried M, Bennouna J, Bondarenko I, Douillard JY, Heigener DF, Krzakowski M, Mellemgaard A, Novello S, Orlov S, Summers Y, von Pawel J, Stohr J, Kaiser R, Reck M. Efficacy and Safety of Nintedanib Plus Docetaxel in Patients with Advanced Lung Adenocarcinoma: Complementary and Exploratory Analyses of the Phase III LUME-Lung 1 Study. Target Oncol. 2017 Aug;12(4):475-485. doi: 10.1007/s11523-017-0517-2. PMID 28702806
- [Derived] Reck M, Kaiser R, Mellemgaard A, Douillard JY, Orlov S, Krzakowski M, von Pawel J, Gottfried M, Bondarenko I, Liao M, Gann CN, Barrueco J, Gaschler-Markefski B, Novello S; LUME-Lung 1 Study Group. Docetaxel plus nintedanib versus docetaxel plus placebo in patients with previously treated non-small-cell lung cancer (LUME-Lung 1): a phase 3, double-blind, randomised controlled trial. Lancet Oncol. 2014 Feb;15(2):143-55. doi: 10.1016/S1470-2045(13)70586-2. Epub 2014 Jan 9. PMID 24411639

RESULTS

PARTICIPANT FLOW:
Groups:
- Nintedanib Plus Docetaxel: Nintedanib 200 mg twice daily administered orally in the form of a soft gelatin capsule plus docetaxel 75 milligram (mg)/square meter (m2) once every 3 weeks administered via intravenous infusion over 1 hour (h).
- Placebo Plus Docetaxel: Placebo soft gelatin capsule matching that of nintedanib 2 times daily plus docetaxel 75 mg/m2 once every 3 weeks administered via intravenous infusion over 1 hour (h).
Period: Overall Study
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Started | 655 (randomised patients) | 659 (randomised patients)
Completed | 6 | 5
Not Completed | 649 | 654
Not completed — Progressive disease (modified RECIST) | 404 | 435
Not completed — Worsening or AE of underlying disease | 64 | 70
Not completed — Other AE | 84 | 73
Not completed — Protocol Violation | 9 | 9
Not completed — Lost to Follow-up | 5 | 5
Not completed — Withdrawal by Subject | 60 | 42
Not completed — Not treated | 3 | 4
Not completed — Reasons other than stated above | 20 | 16

BASELINE CHARACTERISTICS:
Population: Randomised Set (RS)- Includes all randomised patients, whether patients had received study treatment or not
Groups:
- Total: Total of all reporting groups
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel | Total
Number analyzed (Participants) | 655 | 659 | 1314
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (9.7) | 59.8 (9.0) | 59.7 (9.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 179 | 180 | 359
  Male | 476 | 479 | 955
Tumour histology [Count of Participants; unit: Participants]
  Adenocarcinoma | 322 | 336 | 658
  Squamous cell carcinoma | 276 | 279 | 555
  Other | 57 | 44 | 101
Number of patients with adenocarcinoma and time since first line therapy in categories [Count of Participants; unit: Participants] — Population: Randomised patients with adenocarcinoma and time since first line therapy.
  Participants
    number analyzed (Participants) | 322 | 336 | 658
    <9 month | 206 | 199 | 405
    >=9 month | 112 | 134 | 246
    Missing | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) as Assessed by Central Independent Review
Description: Progression Free Survival (PFS) as assessed by central independent review according to the modified Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) . Progression free survival (PFS) is defined as the duration of time from date of randomisation to date of progression or death (whatever occurs earlier).
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until cut-off date 2 November 2010 (when 713 PFS events were observed)
Population: Randomised Set
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 565 | 569
months | 3.4 [1.5 to 5.7] | 2.7 [1.4 to 4.6]
Statistical Analysis 1: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; HR, Confidence Interval (CI) and p-value obtained from the proportional hazards model stratified by baseline ECOG PS (0 vs 1), tumour histology (squamous vs non-squamous), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Test type: Superiority or Other; p = 0.0019, Regression, Cox; Hazard Ratio (HR) = 0.79, 95% CI 2-sided [0.68 to 0.92] — Hazard Ratio (HR) below 1 favors nintedanib

2. Secondary Outcome: Overall Survival (Key Secondary Endpoint)
Description: Overall Survival (OS) defined as the duration from randomisation to death (irrespective of the reason of death). Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
  A fixed-sequence-testing was implemented for key secondary endpoint if both the primary and the follow-up analysis showed a treatment benefit (P<0.05) of nintedanib over placebo. In this case, the OS would be tested using hierarchical testing of statistical hypotheses in (1) patients with adenocarcinoma and <9 months since start of first-line therapy, (2) patients with adenocarcinoma, and (3) all patients. Each hypothesis could be only tested at the pre-specified alpha level if the previous null hypothesis in the testing sequence had been.
Time Frame: From randomisation until cut-off date 15 February 2013 (approximately 48 months or 1151 deaths among all patients )
Population: Randomised Set
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
months
  Adenocarcinoma and <9 months: number analyzed (Participants) | 206 | 199
  Adenocarcinoma and <9 months | 10.9 [5.1 to 21.9] | 7.9 [4.5 to 14.5]
  Adenocarcinoma: number analyzed (Participants) | 322 | 336
  Adenocarcinoma | 12.6 [5.5 to 24.2] | 10.3 [5.5 to 19.9]
  All patients | 10.1 [5.0 to 19.4] | 9.1 [4.8 to 17.2]
Statistical Analysis 1: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Hierarchical testing was tested in a fixed sequence of statistical hypotheses in (1) patients with adenocarcinoma and <9 months since start of first-line therapy, (2) patients with adenocarcinoma, and (3) all patients. Each hypothesis could be only tested at the pre-specified alpha level if the previous null hypothesis in the testing sequence had been rejected. Overall survival for patients with adenocarcinoma and <9 months since start of first line therapy; Test type: Superiority or Other; p = 0.0073, Regression, Cox — HR, CI and p-value obtained from the prop. hazards model stratified by baseline ECOG PS (0 vs 1 - one pat. had 2), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.60 to 0.92] — The overall alpha level followed a Lan-DeMets spending function with O'Brien-Fleming shape parameter to preserve an overall 2-sided alpha level of 0.05. HR below 1 favors nintedanib
Statistical Analysis 2: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Hierarchical testing was tested in a fixed sequence of statistical hypotheses in (1) patients with adenocarcinoma and <9 months since start of first-line therapy, (2) patients with adenocarcinoma, and (3) all patients. Each hypothesis could be only tested at the pre-specified alpha level if the previous null hypothesis in the testing sequence had been rejected. Overall survival for patients with adenocarcinoma; Test type: Superiority or Other; p = 0.0359, Regression, Cox — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.83, 95% CI 2-sided [0.70 to 0.99] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Hierarchical testing was tested in a fixed sequence of statistical hypotheses in (1) patients with adenocarcinoma and <9 months since start of first-line therapy, (2) patients with adenocarcinoma, and (3) all patients. Each hypothesis could be only tested at the pre-specified alpha level if the previous null hypothesis in the testing sequence had been rejected. Overall survival for all patients; Test type: Superiority or Other; p = 0.2720, Regression, Cox — HR, CI and p-value obtained from the prop. hazards model stratified by baseline ECOG PS (0 vs 1 - one pat. had 2), tumour histology (squamous vs non-squamous), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Hazard Ratio (HR) = 0.94, 95% CI 2-sided [0.83 to 1.05] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Follow-up Analysis of Progression Free Survival (PFS) as Assessed by Central Independent Review
Description: Follow-up analysis was conducted at the time of overall survival analysis. Progression Free Survival (PFS) as assessed by central independent review according to the modified RECIST (version 1.0) criteria.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised Set
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Nintedanib Plus Docetaxel: Nintedanib 200 mg twice daily administered orally in a form of a soft gelatin capsule plus docetaxel 75 mg/m2 once every 3 weeks administered via intravenous infusion over 1 hour (h).
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
months | 3.5 [1.5 to 5.7] | 2.7 [1.4 to 5.5]
Statistical Analysis 1: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Test type: Superiority or Other; p = 0.0070, Regression, Cox — HR, CI and p-value obtained from the proportional hazards model stratified by baseline ECOG PS (0 vs 1), tumour histology (squamous vs non-squamous), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.75 to 0.96] — HR below 1 favors nintedanib

4. Secondary Outcome: Follow-up Analysis of Progression Free Survival (PFS) as Assessed by Investigator
Description: Follow-up analysis was conducted at the time of overall survival analysis. Progression Free Survival (PFS) as assessed by investigator according to the modified RECIST (version 1.0) criteria.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised Set
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
months | 4.2 [2.1 to 7.1] | 3.0 [1.4 to 5.7]
Statistical Analysis 1: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Test type: Superiority or Other; p = 0.0012, Regression, Cox — [p-value comment as in outcome 3, analysis 1]; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.73 to 0.93] — HR below 1 favors nintedanib

5. Secondary Outcome: Objective Tumour Response
Description: Confirmed objective response is defined as confirmed Complete Response (CR) and Partial Response (PR) and evaluated according to the modified RECIST criteria version 1.0.
  As per RECIST v1.0, Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised Set
Measure: Number; unit: % of participants
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
% of participants
  central independent reviewer | 4.4 | 3.3
  investigator assessment | 10.4 | 7.6
Statistical Analysis 1: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Analysis based on the central independent review; Test type: Superiority or Other; p = 0.3067, Regression, Logistic — Odds ratio and p-value are obtained from logistic regression model adjusted for baseline ECOG PS (0 vs 1); Odds Ratio (OR) = 1.34, 95% CI 2-sided [0.76 to 2.39] — An odds ratio >1 indicates a benefit to nintedanib
Statistical Analysis 2: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Analysis based on the investigator's assessment; Test type: Superiority or Other; p = 0.0761, Regression, Logistic — Odds ratio and p-value are obtained from logistic regression model adjusted for baseline ECOG PS (0 vs 1); Odds Ratio (OR) = 1.41, 95% CI 2-sided [0.96 to 2.08] — An odds ratio >1 indicates a benefit to nintedanib

6. Secondary Outcome: Duration of Confirmed Objective Tumour Response
Description: The duration of objective response is the time from first documented (CR) or (PR) to the time of progression or death and evaluated according to the modified RECIST criteria version 1.0.
  As per RECIST v1.0, Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised Set
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
months
  central independent reviewer: number analyzed (Participants) | 29 | 22
  central independent reviewer | 4.3 [3.0 to 5.7] | 4.3 [2.8 to 8.5]
  investigator assessment: number analyzed (Participants) | 68 | 50
  investigator assessment | 5.7 [4.1 to 10.0] | 5.5 [3.9 to 9.6]

7. Secondary Outcome: Time to Confirmed Objective Tumour Response
Description: Time to confirmed objective response is defined as time from randomisation to the date of first documented (CR) or (PR) and evaluated according to the modified RECIST criteria version 1.0.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised Set
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
months
  central independent reviewer: number analyzed (Participants) | 29 | 22
  central independent reviewer | 1.5 [1.4 to 3.0] | 2.9 [1.4 to 5.6]
  investigator assessment: number analyzed (Participants) | 68 | 50
  investigator assessment | 2.6 [1.4 to 4.0] | 2.7 [1.4 to 4.1]

8. Secondary Outcome: Disease Control
Description: Disease control was defined as a best overall response of Complete Response (CR), Partial Response (PR), or Stable Disease (SD) and evaluated according to the modified RECIST criteria version 1.0.
  As per RECIST v1.0 for target lesions : Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression.
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised Set
Measure: Number; unit: % of participants
Groups:
- Placebo Plus Docetaxel: Placebo soft gelatin capsule matching that of nintedanib 2 times daily plus docetaxel 75 mg/m2 (with dose reduction to 60 mg/m2 if required) once every 3 weeks administered via intravenous infusion over 1 hour (h).
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
% of participants
  central independent reviewer: number analyzed (Participants) | 354 | 272
  central independent reviewer | 54.0 | 41.3
  investigator assessment: number analyzed (Participants) | 415 | 339
  investigator assessment | 63.4 | 51.4
Statistical Analysis 1: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Analysis based on the central independent review; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Odds ratio and p-value are obtained from logistic regression model adjusted for baseline ECOG PS (0 vs 1); Odds Ratio (OR) = 1.68, 95% CI 2-sided [1.35 to 2.09] — An odds ratio >1 indicates a benefit to nintedanib
Statistical Analysis 2: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Analysis based on investigator's assessment; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — Odds ratio and p-value are obtained from logistic regression model adjusted for baseline ECOG PS (0 vs 1); Odds Ratio (OR) = 1.64, 95% CI 2-sided [1.31 to 2.05] — An odds ratio >1 indicates a benefit to nintedanib

9. Secondary Outcome: Duration of Disease Control
Description: The duration of disease control was defined as the time from randomisation to the date of disease progression or death (which ever occurs first) for patients with disease control.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised Set
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
months
  central independent reviewer: number analyzed (Participants) | 354 | 272
  central independent reviewer | 5.6 [4.1 to 7.1] | 5.6 [4.0 to 8.2]
  investigator assessment: number analyzed (Participants) | 415 | 339
  investigator assessment | 5.7 [4.2 to 8.4] | 5.6 [4.1 to 8.5]

10. Secondary Outcome: Change From Baseline in Tumour Size
Description: Percentage change from baseline in tumour size is defined as decrease in the sum of the longest diameter of the target lesion.
  Presented means are in fact adjusted best means percentage changes generated from ANOVA model adjusted for baseline ECOG PS (0 vs. 1), tumour histology (squamous vs non-squamous), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no)
  This endpoint was analysed based on the central independent reviewer as well as the investigator.
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised Set
Measure: Mean (95% Confidence Interval); unit: percentage of change in tumor size in mm
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
percentage of change in tumor size in mm
  central independent reviewer: number analyzed (Participants) | 582 | 570
  central independent reviewer | -4.87 [-6.62 to -3.12] | 0.58 [-1.19 to 2.35]
  investigator assessment: number analyzed (Participants) | 603 | 596
  investigator assessment | -10.34 [-12.58 to -8.11] | -2.14 [-4.39 to 0.10]
Statistical Analysis 1: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Analysis based on the central independent review; Test type: Superiority or Other; p < 0.0001, ANOVA — P-value generated from ANOVA model adjusted for baseline ECOG PS (0 vs. 1), tumour histology (squamous vs non-squamous), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no)
Statistical Analysis 2: Comparison: Nintedanib Plus Docetaxel vs Placebo Plus Docetaxel; Analysis based on the investigator's assessment; Test type: Superiority or Other; p < 0.0001, ANOVA — [p-value comment as in outcome 10, analysis 1]

11. Secondary Outcome: Clinical Improvement
Description: Clinical improvement was defined as the time from randomisation to deterioration in body weight and/or Eastern Cooperative Oncology group performance score (ECOG PS) whichever occurred first.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve.
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised set
Measure: Median (Inter-Quartile Range); unit: months
Groups:
- Nitedanib Plus Docetaxel: Nintedanib 200 mg twice daily administered orally in a form of a soft gelatin capsule plus docetaxel 75 mg/m2 once every 3 weeks administered via intravenous infusion over 1 hour (h).
Arm/Group | Nitedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
months | 5.9 [2.1 to 22.7] | 5.2 [2.1 to 19.2]
Statistical Analysis 1: Comparison: Nitedanib Plus Docetaxel vs Placebo Plus Docetaxel; Test type: Superiority or Other; p = 0.7282, Regression, Cox — HR, CI and p-value obtained from the prop. hazards model stratified by baseline ECOG PS (0 vs 1 - one pat.had 2), tumour histology (squamous vs non-squamous), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Hazard Ratio (HR) = 1.03, 95% CI 2-sided [0.87 to 1.21] — HR below 1 favors nintedanib

12. Secondary Outcome: Quality of Life (QoL)
Description: Quality of life (QoL) was measured by standardised questionnaires (Health Status Self-Assessment Questionnaire (EQ-5D), EORTC Quality of life questionnaire - Core 30 (EORTC QLQ-C30), Quality of life questionnaire - lung cancer module (EORTC QLQ-LC13). The EORTC QLQ-C30 comprises of 30 questions, using both multi-item scales and single-item measures. EORTC LC-13 comprises of 13 questions incorporating 1 multi-item scale and a series of single items.
  The following were the main points of interest:
  Time to deterioration of cough (EORTC QLQ-LC13 question 1), Time to deterioration of dyspnoea (QLQ-LC13, composite of questions 3 to 5), Time to deterioration of pain (QLQ- C30, composite of questions 9 and 19).
  Time to deterioration of cough, dyspnoea and pain was defined as the time to a 10-point increase from the baseline score.
  Median, 25th and 75th percentiles are calculated from an unadjusted Kaplan-Meier curve
Time Frame: From randomisation until cut-off date 15 February 2013
Population: Randomised set
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Nitedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 655 | 659
months
  Time to deterioration of cough | 4.3 [1.6 to 11.8] | 3.5 [1.5 to 12.6]
  Time to deterioration of dyspnoea | 2.0 [0.8 to 4.2] | 2.1 [0.8 to 4.5]
  Time to deterioration of pain | 2.8 [1.1 to 6.5] | 2.6 [0.8 to 5.8]
Statistical Analysis 1: Comparison: Nitedanib Plus Docetaxel vs Placebo Plus Docetaxel; Analysis evaluating the time to deterioration of cough; Test type: Superiority or Other; p = 0.1858, Regression, Cox — HR, CI and p-value obtained from the prop. hazards model stratified by baseline ECOG PS (0 vs >=1), tumour histology (squamous vs non-squamous), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Hazard Ratio (HR) = 0.90, 95% CI 2-sided [0.77 to 1.05] — HR below 1 favors nintedanib
Statistical Analysis 2: Comparison: Nitedanib Plus Docetaxel vs Placebo Plus Docetaxel; Analysis evaluating the time to deterioration of dyspnoea; Test type: Superiority or Other; p = 0.5203, Regression, Cox — [p-value comment as in outcome 12, analysis 1]; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.91 to 1.20] — HR below 1 favors nintedanib
Statistical Analysis 3: Comparison: Nitedanib Plus Docetaxel vs Placebo Plus Docetaxel; Analysis evaluating the time to deterioration of pain; Test type: Superiority or Other; p = 0.4373, Regression, Cox — HR, CI and p-value obtained from the prop. hazards model stratified by baseline ECOG PS (0 vs >= 1), tumour histology (squamous vs non-squamous), brain metastases at baseline (yes vs no) and prior treatment with bevacizumab (yes vs no); Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.82 to 1.09] — HR below 1 favors nintedanib

13. Secondary Outcome: Dose Normalised Predose Plasma Concentration at Steady State (Cpre,ss,Norm) of Nintedanib and of Its Metabolites BIBF 1202 and BIBF 1202 Glucuronide
Description: Geometric mean of dose normalised predose plasma concentration (Cpre,ss,norm) of nintedanib and of its metabolites BIBF 1202 and BIBF 1202 glucuronide evaluated at steady state based on course 2 and 3. If only one value was available and valid, then this value was used for calculation of Cpre,ss,norm.
Time Frame: Before the administration of nintedanib or placebo and between a window of 30 mins to an hour after administration of trial drug during Course 2 and between 1 and 3 hours after administration of trial drug during Course 3
Population: Pharmacokinetic set- all patients in the treated set who were documented to have received at least 1 dose of nintedanib and who had at least 1 valid drug plasma concentration available
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL/mg
Groups:
- Nitedanib 200 mg Bid Plus Docetaxel: Nintedanib 200 mg twice daily administered orally in a form of a soft gelatin capsule plus docetaxel 75 mg/m2 once every 3 weeks administered via intravenous infusion over 1 hour (h).
- Nintedanib 150 Bid mg Plus Docetaxel: Nintedanib 150 mg twice daily administered orally in a form of a soft gelatin capsule plus docetaxel 75 mg/m2 once every 3 weeks administered via intravenous infusion over 1 hour (h).
Arm/Group | Nitedanib 200 mg Bid Plus Docetaxel | Nintedanib 150 Bid mg Plus Docetaxel
Number analyzed (Participants) | 454 | 38
ng/mL/mg
  nintedanib: number analyzed (Participants) | 453 | 38
  nintedanib | 0.0707 (77.7) | 0.106 (52.6)
  metabolite BIBF 1202 | 0.0907 (127) | 0.190 (152)
  metabolite BIBF 1202 glucuronide: number analyzed (Participants) | 429 | 33
  metabolite BIBF 1202 glucuronide | 1.04 (153) | 1.94 (135)

14. Secondary Outcome: Incidence and Intensity of Adverse Events
Description: Incidence and intensity of adverse events according to the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. The worst CTCAE grade per patient is reported and MedDRA version 15.1 used.
  Serious signs and symptoms of progressive disease were reported as an adverse event in analysis of this endpoint.
Time Frame: From the first drug administration until 28 days after the last drug administration, up to 42 months
Population: Treated set- all randomised patients who were documented to have taken at least 1 dose of study medication . Patients were allocated to the treatment groups according to the treatment actually received.
Measure: Number; unit: % of participants
Arm/Group | Nitedanib Plus Docetaxel | Placebo Plus Docetaxel
Number analyzed (Participants) | 652 | 655
% of participants
  Grade 1 | 5.7 | 8.2
  Grade 2 | 16.6 | 20.5
  Grade 3 | 21.2 | 21.2
  Grade 4 | 33.7 | 31.3
  Grade 5 | 16.4 | 11.8

ADVERSE EVENTS:
Time Frame: From the first drug administration until 28 days after the last drug administration, up to 42 months
Description: Number of participants at risk corresponds to all randomised patients who were documented to have taken at least 1 dose of study medication. Patients were allocated to the treatment groups according to the treatment actually received.
Arm/Group | Nintedanib Plus Docetaxel | Placebo Plus Docetaxel
All-Cause Mortality (participants affected / at risk) | 107/652 | 77/655
Serious Adverse Events (participants affected / at risk) | 224/652 | 206/655
Other Adverse Events (participants affected / at risk) | 569/652 | 547/655
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib Plus Docetaxel (N=652) | Placebo Plus Docetaxel (N=655)
Anaemia (Blood and lymphatic system disorders) | 2 | 6
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 30 | 19
Leukopenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 21 | 21
Pancytopenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 2
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 5 | 2
Atrial flutter (Cardiac disorders) | 1 | 2
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 2
Cardio-respiratory arrest (Cardiac disorders) | 1 | 2
Cardiopulmonary failure (Cardiac disorders) | 1 | 2
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 3
Pericardial effusion (Cardiac disorders) | 4 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Tachyarrhythmia (Cardiac disorders) | 2 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 2
Diplopia (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 16 | 13
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 0 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Neutropenic colitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 3
Vomiting (Gastrointestinal disorders) | 8 | 7
Asthenia (General disorders) | 7 | 4
Chest discomfort (General disorders) | 1 | 1
Chest pain (General disorders) | 7 | 8
Condition aggravated (General disorders) | 1 | 0
Death (General disorders) | 2 | 1
Device occlusion (General disorders) | 0 | 1
Extravasation (General disorders) | 0 | 1
Fatigue (General disorders) | 7 | 1
Feeling abnormal (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 11 | 8
Malaise (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 1
Multi-organ failure (General disorders) | 2 | 1
Oedema peripheral (General disorders) | 1 | 0
Organ failure (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Performance status decreased (General disorders) | 1 | 0
Pyrexia (General disorders) | 7 | 9
Bile duct obstruction (Hepatobiliary disorders) | 1 | 1
Cholecystocholangitis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 2 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 2
Hypersensitivity (Immune system disorders) | 0 | 3
Abscess rupture (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 4
Bronchopneumonia (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Empyema (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 1 | 0
Febrile infection (Infections and infestations) | 0 | 1
Folliculitis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Gastrointestinal infection (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 2
Infectious pleural effusion (Infections and infestations) | 2 | 1
Influenza (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 4 | 3
Lung abscess (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Neutropenic infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Opportunistic infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 17 | 26
Pulmonary tuberculosis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 3
Respiratory tract infection bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 7 | 3
Septic shock (Infections and infestations) | 2 | 0
Streptococcal infection (Infections and infestations) | 0 | 1
Tuberculosis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 3
Urinary tract infection (Infections and infestations) | 1 | 2
Acetabulum fracture (Injury, poisoning and procedural complications) | 0 | 1
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 1
Haemoglobin decreased (Investigations) | 3 | 2
Hepatic enzyme increased (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 0 | 1
Neutrophil count decreased (Investigations) | 6 | 3
Weight decreased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1
Hepatic cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 25 | 17
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Metastases to chest wall (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Aphasia (Nervous system disorders) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 2
Cerebral infarction (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Cognitive disorder (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 4 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Diplegia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 2
Encephalopathy (Nervous system disorders) | 0 | 1
Epiduritis (Nervous system disorders) | 0 | 1
Facial paresis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intracranial pressure increased (Nervous system disorders) | 1 | 2
Ischaemic stroke (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0
Loss of consciousness (Nervous system disorders) | 2 | 0
Monoparesis (Nervous system disorders) | 0 | 1
Nervous system disorder (Nervous system disorders) | 0 | 1
Neuralgia (Nervous system disorders) | 1 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Paraparesis (Nervous system disorders) | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Confusional state (Psychiatric disorders) | 0 | 2
Depression (Psychiatric disorders) | 4 | 0
Disorientation (Psychiatric disorders) | 0 | 3
Mental disorder due to a general medical condition (Psychiatric disorders) | 1 | 1
Panic attack (Psychiatric disorders) | 1 | 0
Personality change (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 2
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Alveolitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Bronchial haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bronchial secretion retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchostenosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 | 30
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 6 | 7
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 8 | 8
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 6
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 5 | 3
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 | 2
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 1
Haemorrhage (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 3 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1
Subclavian artery thrombosis (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 1 | 1
Thrombosis (Vascular disorders) | 0 | 1
Venous thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis limb (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nintedanib Plus Docetaxel (N=652) | Placebo Plus Docetaxel (N=655)
Anaemia (Blood and lymphatic system disorders) | 33 | 43
Neutropenia (Blood and lymphatic system disorders) | 69 | 73
Abdominal pain (Gastrointestinal disorders) | 35 | 37
Constipation (Gastrointestinal disorders) | 35 | 76
Diarrhoea (Gastrointestinal disorders) | 260 | 130
Nausea (Gastrointestinal disorders) | 158 | 117
Stomatitis (Gastrointestinal disorders) | 62 | 54
Vomiting (Gastrointestinal disorders) | 102 | 54
Asthenia (General disorders) | 51 | 60
Chest pain (General disorders) | 49 | 54
Fatigue (General disorders) | 191 | 175
Oedema peripheral (General disorders) | 35 | 42
Pyrexia (General disorders) | 76 | 89
Alanine aminotransferase increased (Investigations) | 184 | 55
Aspartate aminotransferase increased (Investigations) | 145 | 43
Blood alkaline phosphatase increased (Investigations) | 38 | 9
Haemoglobin decreased (Investigations) | 70 | 77
Neutrophil count decreased (Investigations) | 236 | 232
White blood cell count decreased (Investigations) | 157 | 158
Decreased appetite (Metabolism and nutrition disorders) | 144 | 101
Arthralgia (Musculoskeletal and connective tissue disorders) | 40 | 46
Back pain (Musculoskeletal and connective tissue disorders) | 26 | 44
Myalgia (Musculoskeletal and connective tissue disorders) | 40 | 45
Pain in extremity (Musculoskeletal and connective tissue disorders) | 31 | 41
Dizziness (Nervous system disorders) | 31 | 34
Dysgeusia (Nervous system disorders) | 31 | 34
Headache (Nervous system disorders) | 39 | 42
Peripheral sensory neuropathy (Nervous system disorders) | 40 | 47
Insomnia (Psychiatric disorders) | 31 | 38
Cough (Respiratory, thoracic and mediastinal disorders) | 96 | 108
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 100 | 80
Alopecia (Skin and subcutaneous tissue disorders) | 107 | 119

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.